CLINICAL TRIAL: NCT00177021
Title: Aldara for the Treatment of Extensive Alopecia Areata
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hordinsky, Maria K., MD (Individual)
Collaborators: National Alopecia Areata Foundation (Other); 3M (Industry)
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9908M15841
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-11-13 (Estimated); Status verified 2006-11

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

INTERVENTIONS:
Drug: Aldara Cream 5%

SUMMARY:
We propose to examine the efficacy and tolerability of Aldara Cream 5% for the treatment of extensive alopecia areata. Aldara is a immune-response modifier. The drug induces the production of cytokines which are small, hormone-like proteins involved in cellular communication during immune responses. We hypothesize that this drug will effect the inflammatory cells present around hair follicles in patients with alopecia areata.

DETAILED DESCRIPTION:
Ten patients with extensive scalp alopecia areata (>95% hair loss)of less than 2 years duration will be invited to participate in this study. For six months each person will be asked to apply Aldara Cream 5% daily to the right half of the scalp. No drug will be applied to the left side. Skin biopsies will be taken of the right scalp before and at the completion of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Must be 18 years of age, male or female of any race.
* Subjects must have extensive scalp alopecia areata (>95% involvement) of less than 2 years duration.
* In good general and mental health based on a medical history and physical exam.
* Patient must be willing to refrain from all other alopecia areata treatments during the course of the study.
* Must agree to shampoo daily with Free and Clear shampoo.

Exclusion Criteria:

* History of any illness or condition that in the opinion of the investigator might confound the results of the study or pose additional risk in administering the drug to the patient.
* Significant abnormalities on screening clinical examination.
* Previous use of Aldara Cream 5%
* History of drug or alcohol abuse.
* Use of ultraviolet radiation, including tanning beds and PUVA therapy for treatment of acne, psoriasis, or any other skin condition within 2 months prior to study initiation.
* Use of systemic or topical glucocorticoids, corticosteroids. estrogenic, progestogenic, androgenic, or antiandrogen drugs, cyclosporine, FK506 or immunotherapy with DNCB, SADBE, or DCP within 6 months of study initiation.
* Use of a topical medication within six weeks prior to the study.
* Alterations in thyroid medication within 6 months of study initiation.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2000-10; Study Completion 2002-08

PRIMARY OUTCOMES:
To determine the efficacy of Aldara Cream 5% for the treatment of extensive alopecia areata

SECONDARY OUTCOMES:
Assess changes in the hair follicle differentiation oand perifollicular inflammation before and after treatment with Aldara Cream5%

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Marna Ericson, Ph D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States